CLINICAL TRIAL: NCT05760521
Title: Optimizing Rural Community Health Through Interdisciplinary Dementia Detection and Care
Brief Title: Optimizing Rural Community Health Through Dementia Detection and Care
Acronym: ORCHID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Atlantic University (Other)
Collaborators: University of Miami (Other); Palm Beach State College (Unknown)
Responsible Party: Principal Investigator, Lisa A Wiese, Associate Professor, Nursing, Florida Atlantic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1851318
Record Dates: First submitted 2023-01-24; First posted 2023-03-08 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Alzheimer' Disease
Keywords: Rural; Multicultural; Early Detection; Multidisciplinary
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will not know to which Randomized group that they have been assigned (intervention or control).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Provider Educational Intervention (Experimental): Providers receiving education/support from neurology teams, Adult Gerontological Nurse Practitioner (AGNP) assessments/recommendations, and training of office staff regarding ADRD and community resources support for patients/caregivers.
  Interventions: Other: Provider Educational Intervention
- Arm B: Provider Control (No Intervention): Providers receiving AGNP assessments/recommendations only.

INTERVENTIONS:
Other: Provider Educational Intervention — Following the informed consent (10 min) and sociodemographic survey (5 minutes), the providers in Arm A will be offered education of two days, six hours each day, with support and follow-up. They will also be asked to complete brief knowledge and confidence surveys pre-post-intervention (30 minutes total).
  Arms: Arm A: Provider Educational Intervention

SUMMARY:
The overall goal of this one-year study is to test a comprehensive protocol for Alzheimer's Disease and Related Dementias (ADRD) diagnosis and care management that can be used as a model for rural communities, which experience low rates of dementia diagnosis and treatment.

DETAILED DESCRIPTION:
The ORCHID study integrates 1) A one-group community educational intervention focused on increasing community awareness of brain-health promoting behaviors and dementia literacy and knowledge; and 2) A primary care provider dementia educational intervention designed to improve provider knowledge and confidence in detecting, diagnosing, and treating patients with cognitive impairment, with the goal of increasing ADRD diagnosis and treatment rates, reducing dementia-related hospitalization rates, increasing utilization of available local support services, and improving caregiver-related outcomes.

The community education intervention is a 6-week culturally-relevant educational program focused on brain health promotion. Effects of the community intervention on dementia knowledge and literacy will be assessed with a pre-post analytic approach using paired t-tests to compare changes in mean AD knowledge and literacy. The provider dementia educational intervention uses a cluster-randomized trial design with participating primary care provider offices randomly assigned to either receive the intervention (Arm A) or the control group (Arm B). Providers assigned to Arm A receive an educational intervention that includes training in ADRD detection, diagnosis, and care management. Providers assigned to Arm B do not receive educational intervention. Both groups receive the following: detailed reports from neuropsychological testing performed by a study clinician, hands-on training of provider office staff on dementia screening tools, and support with referrals to local support services. The two study groups (Arms A and B) will be compared on: 1) change in provider dementia knowledge and confidence, caregiver burden and self-efficacy; and 2) rates of dementia diagnosis and treatment, rates of dementia-related hospital admissions, and rates of referral to support service. A generalized linear mixed model analytic approach will be used to assess the effect of the provider intervention on study outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years and older
* Lives in the Glades Area of Florida
* Lives in the community/ be non-institutionalized
* Has no known diagnosis of Alzheimer's Disease and Related Dementias
* Speaks either English, Spanish, or Creole
* Has no known plans to move out of the Glades Area in the next 12 months

Exclusion Criteria:

* Previous diagnosis of a dementia-related illness
* Aged under 50 years

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change in rates of new dementia diagnosis and treatment | at baseline, 3 months, 6 months, and 12 months post-intervention
  The intervention and control groups will be compared on rates of dementia diagnosis and treatment at four different time points; baseline and post-intervention.
Change in rates of referrals to Area Support Services | baseline, 3 months, 6 months, and 12 months post-intervention
  The intervention and control groups will be compared on rates of referrals to support service at four different time points; baseline and post-intervention.
Change in AD knowledge | : 6 weeks
  Alzheimer's Disease Knowledge Scale (ADKS) will be collected from participants in the community educational intervention before (week 0) and immediately after the intervention (week 6). Scores on the ADKS range from 0 to 13, with higher scores indicating greater knowledge
Change in AD literacy treatment plan. | 6 weeks
  Dementia Literacy Assessment (DELA) will be administered as part of the community educational intervention before (week 0) and immediately after the intervention (week 6). DELA consists of 25 items scored 0=incorrect/1=correct. Total DELA score ranges from 0 to 25 with a higher score being indicative of greater dementia literacy.

SECONDARY OUTCOMES:
Change in rates of preventable admission related to ADRD to the local hospital | at baseline, 3 months, and 6 months post-intervention
  The intervention and control groups will be compared on rates of hospitalization for ADRD-related complications, at baseline and at three different time points post-intervention.
Change in provider knowledge related to ADRD | at baseline, 3 months, and 6 months post-intervention
  Alzheimer's Disease Knowledge Scale (ADKS) will be administered at baseline, and at three different time points post-intervention.
Change in provider confidence in establishing an ADRD diagnosis and treatment plan | at baseline, 3 months, and 6 months post-intervention
  General Practitioners' Attitude and Confidence Scale for Dementia (GPACS-D) will be administered at baseline, and at three different time points post-intervention, in the intervention and control groups. Total scores range from 15 to 75, with higher scores indicating greater confidence and attitudes towards dementia.
Change in caregiver burden | at baseline, 3 months, and 6 months post-intervention
  The 12-item Zarit Burden Inventory (ZBI) will be collected at baseline, and at three different time points post-intervention, in the intervention and control groups. Scores range from 0 to 48, with higher scores indicating greater burden.
Change in caregiver self-efficacy | at baseline, 3 months, and 6 months post-intervention
  The Revised Scale for Caregiver Self-Efficacy (RSCSE) will be administered at baseline, and at three different time points post-intervention, in the intervention and control groups. RSCSE consists of 3 subscales (Self-Efficacy for Obtaining Respite; Self-Efficacy for Responding to Disruptive Patient Behaviors; and Self-Efficacy for Controlling Upsetting Thoughts about Caregiving), each consisting of 5 statements scored on a 0-100 with higher scores indicating better self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Wiese, Principal Investigator — Florida Atlantic University, C.E. Lynn College of Nursing; Magdalena I Tolea, PhD, Principal Investigator — University of Miami; Joanne Pulido, Principal Investigator — Palm Beach State College
Locations (2):
- United States (2):
  - Palm Beach State College, Belle Glade, Florida
  - Florida Atlantic University, Boca Raton, Florida

IPD SHARING:
Plan to Share IPD: Yes
Data will be de-identified and stored on the PI's university Biomedical Health Research Informatics Core (BHRIC) which is an isolated and independently secured infrastructure managed by the FAU Office of Information technology. The BHRIC Data managed system includes limited access controls, software firewalls, and network-wide virus protection, and daily backups. Data export for analysis is expected to be automated export procedures allowing for seamless download of data into Excel or other widely used statistical packages (SPSS, SAS). Data output tables will be password protected and maintained via password protected university computers. Limited information (informed consents) will be maintained on paper, numerically coded, and secured under lock and key access (further described under the "Informed Consents" section.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the data has been analyzed and deidentified. We expect that to be within a year of study closure (March 2024).
Access Criteria: By Request, with approval of Data Management Officer, Research Team, and IRB Officials.